CLINICAL TRIAL: NCT07331792
Title: Comparative Efficacy of Topical 1% Clotrimazole vs Oral Itraconazole in the Treatment of Pityriasis Versicolor
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Combined Military Hospital Abbottabad (Other)
Responsible Party: Principal Investigator, Zaeema Aman, Resisent Dermatology, Combined Military Hospital Abbottabad
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CMH-Atd-ETH-200-Derm-25
Record Dates: First submitted 2025-12-19; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Pityriasis Versicolor
MeSH Terms: conditions — Tinea Versicolor | interventions — Itraconazole

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 1% Clotrimazole (Experimental): topical 1 % clotrimazole twice daily for 2 weeks
  Interventions: Drug: Topical 1 % clotrimazole twice daily 2 weeks
- Itraconazole (Experimental): Oral itraconazole 200mg daily 5 days
  Interventions: Drug: Oral itraconazole 200mg daily for 5 days

INTERVENTIONS:
Drug: Topical 1 % clotrimazole twice daily 2 weeks — Topical 1% clotrimazole twice daily for 2 weeks
  Arms: 1% Clotrimazole
Drug: Oral itraconazole 200mg daily for 5 days — Oral itraconazole 200mg daily for 5 days
  Arms: Itraconazole

SUMMARY:
Comparative efficacy of topical 1% clotrimazole vs oral itraconazole in the treatment of pityriasis versicolor -Randomized control trial

ELIGIBILITY:
Inclusion Criteria:

* Age (15-50 years)
* Both genders
* Sufferers of Pityriasis versicolor ( Determined by scale , erythema and pruritus)

Exclusion Criteria:

* Pt with history of antifungals in last one month
* Pt on immunosuppressants or steroid therapy
* Pregnant and lactating women
* Pt with chronic medical conditions ( Diabetes and hypertension)

Ages: 15 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 86 (Estimated)
Dates: Start 2026-02-02 (Estimated); Primary Completion 2026-05-02 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Percentile efficacy of topical versus oral antifungal in the treatment of pityriasis versicolor | 3 months
  Data analysis will be performed using SPSS version 20. The quantitative variable (age, BMI and duration of PV) will be presented as mean ± standard deviation (SD) or median interquartile range (IQR) after checking normality of data by using Shapiro-Wilk test. Frequency and percentages will be used for categorical variables (gender, severity of PV, area of residence, level of education and efficacy). Efficacy will be compared between groups using Chi-square or Fisher exact test. Efficacy will be stratified by age, gender, BMI, duration of PV and severity of PV to deal with effect modifiers. Post-stratification chi-square test or Fischer exact test will be used as test of significance. A p-value of ≤ 0.05 will be considered statistically significant.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bamford JTM, Flores-GenuinoRNS, Ray S, Bigby M, Morales-Sánchez MA, Arkoncel M, et al. Interventions for the treatment of pityriasis versicolor. Cochrane Database Syst Rev. 2018;2018(6):CD011208. https://doi.org/10.1002/14651858.CD011208.pub2
- [Background] Hill RC, Faria W, Gold JAW, Lipner SR. Factors associated with pityriasis versicolor in a large national database. Mycoses. 2024 Aug;67(8):e13775. doi: 10.1111/myc.13775. PMID 39079943
- [Background] Kurniadi I, Hendra Wijaya W, Timotius KH. Malassezia virulence factors and their role in dermatological disorders. Acta Dermatovenerol Alp Pannonica Adriat. 2022 Jun;31(2):65-70. PMID 35751534
- [Background] Leung AK, Barankin B, Lam JM, Leong KF, Hon KL. Tinea versicolor: an updated review. Drugs Context. 2022 Nov 14;11:2022-9-2. doi: 10.7573/dic.2022-9-2. eCollection 2022. PMID 36452877
- [Background] Labedz N, Navarrete-Dechent C, Kubisiak-Rzepczyk H, Bowszyc-Dmochowska M, Pogorzelska-Antkowiak A, Pietkiewicz P. Pityriasis Versicolor-A Narrative Review on the Diagnosis and Management. Life (Basel). 2023 Oct 22;13(10):2097. doi: 10.3390/life13102097. PMID 37895478